CLINICAL TRIAL: NCT05988502
Title: Auricular Acupressure Relieves Constipation for Patients With Heart Failure in Hospital: a Randomised Controlled Trial
Brief Title: Auricular Acupressure Relieves Constipation for Patients With Heart Failure in Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 110269-F
Record Dates: First submitted 2023-07-16; First posted 2023-08-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure; Auricular Acupressure; Constipation; Quality of Life; Depression, Anxiety
Keywords: Anxiety; auricular acupressure; constipation; heart failure; quality of life; Depression
MeSH Terms: conditions — Heart Failure; Constipation; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The participants were randomized into two groups by a research team not involved in the study intervention or data collection. The randomization process was accomplished through a computer-generated sequence of random numbers, and permuted block randomization was employed with four in each block. The random sequence of numbers was separately and sequentially stored in sealed, opaque envelopes that were opened in front of the participants in the predetermined order, which determined their group allocation.the auricular acupressure (AA) group was given auricular acupressure for two weeks and the control group received usual care for heart failure during the same study period. Data were collected consisted of three repeated measurement time points at baseline, Week 1, and Week 2.
Who Masked: Participant, Outcomes Assessor
Masking Description: The random sequence of numbers was separately and sequentially stored in sealed, opaque envelopes that were opened in front of the participants in the predetermined order, which determined their group.The participants do not know their own group, the researcher knows the participant's group and intervenes according to the participant's group, and the outcomes Assessor conducts the outcomes assessment without knowing the participant's group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- auricular acupressure (AA) group (Experimental): the auricular acupressure (AA) group was given auricular acupressure for two weeks
  Interventions: Other: auricular acupressure
- control group (No Intervention): all participants received the same routine care which was general heart failure care and medications for constipation therapy provided by the study hospital professionals. Prior to the study, every participant was assessed by the cardiologist and identified as being appropriate and safe.

INTERVENTIONS:
Other: auricular acupressure — The well-trained researcher nurse in this study was performed the AA intervention. First of all, the participant was instructed to find a comfortable position. Disinfect the ears using cotton with 75 % alcohol was then provided and followed by placed vaccaria seeds (Beijing, China) with an adhesive patch onto the unilateral each selected auricular acupoint (left ear first) Participants were pressed each acupoint by thumb and index finger for one minute, four times a day, five days a week, remove the taped seeds on the 6th day, and then replaced the opposite ear two days after. They were noted that they experienced various sensations while pressing, including numbness, swelling, mild pain, or warmth. Seeds were taped on the other side of the ear weekly for two weeks.
  Two TCM physicians verified the conduct of the AA protocol, which consisted of a selection of acupoints, length of stimulation time, finding location of acupoint, and procedure of practice.
  Arms: auricular acupressure (AA) group

SUMMARY:
This study aimed to investigate the effect of auricular acupressure (AA) to relieve constipation symptoms and improve quality of life in patients hospitalized for their heart failure. A total of 72 participants were randomly assigned and 68 (33 in the AA group and 35 in the control group) completed the study. Outcomes were measured by the Bristolv Stool Form Scale, Constipation Assessment Scale, Patient Assessment of Constipation Symptoms, Visual Scale Analog, Beck Anxiety Inventory and Beck Depression Inventory at baseline, Weeks 1 and 2, as well as Constitution in Chinese Medicine Questionnaire and Patient Assessment of Constipation Quality of Life at baseline and Week 2.

DETAILED DESCRIPTION:
1. Study Design This was a parallel randomized controlled trial with two groups; the auricular acupressure (AA) group was given auricular acupressure for two weeks and the control group received usual care for heart failure during the same study period. Data were collected consisted of three repeated measurement time points at baseline, Week 1, and Week 2.
2. Participants This study consecutively recruited patients who were hospitalized for treating heart failure from the cardiology ward of the a medical center in northern Taiwan. Patients who aged over 20 years and had the New York Heart Association (NYHA) functional classes I-III, constipation(had fewer than three bowel movements a week), and conscious clear and communicable were included, while those who had serious diseases or wounds or infections in both ears were excluded. The sample size required for the study was estimated using G-power software vers.3.1. (Heinrich Heine Universitat, Dusseldorf, Germany), with an effect size of 0.3 referring to the previous study on constipation, the significance level (α) at .05, and 80% statistical power. With considering a 10% dropout rate, a total of 72
3. Randomization and allocation concealment The participants were randomized into two groups by a research team not involved in the study intervention or data collection. The randomization process was accomplished through a computer-generated sequence of random numbers, and permuted block randomization was employed with four in each block. The random sequence of numbers was separately and sequentially stored in sealed, opaque envelopes that were opened in front of the participants in the predetermined order, which determined their group allocation.
4. The auricular acupressure (AA) intervention The AA intervention selected seven acupoints on auricle, including Shenmen (TF4), Intestine (CO7), Rectum (HX2), San Jiao (CO17), Spleen (CO13), Lung (CO14) and Subcortex (AT4), as seen Figure 2 (intestine, rectum, San Jiao, spleen, lung, and subcortex).

   The well-trained researcher nurse in this study was performed the AA intervention. First of all, the participant was instructed to find a comfortable position. Disinfect the ears using cotton with 75 % alcohol was then provided and followed by placed vaccaria seeds (Beijing, China) with an adhesive patch onto the unilateral each selected auricular acupoint (left ear first). Participants were pressed each acupoint by thumb and index finger for one minute, four times a day, five days a week, remove the taped seeds on the 6th day, and then replaced the opposite ear two days after. They were noted that they experienced various sensations while pressing, including numbness, swelling, mild pain, or warmth. Seeds were taped on the other side of the ear weekly for two weeks.

   Two TCM physicians verified the conduct of the AA protocol, which consisted of a selection of acupoints, length of stimulation time, finding location of acupoint, and procedure of practice. In addition, all participants received the same routine care which was general heart failure care and medications for constipation therapy provided by the study hospital professionals. Prior to the study, every participant was assessed by the cardiologist and identified as being appropriate and safe. Data collection was conducted by the same researcher nurse at baseline, Week 1, and Week 2.
5. Measurements Outcomes were assessed by using the Bristolv Stool Form Scale, Constipation Assessment Scale, Patient Assessment of Constipation Symptoms, Visual Scale Analog, Constitution in Chinese Medicine Questionnaire, Beck Anxiety Inventory, Beck Depression Inventory II and Patient Assessment of Constipation Quality Of Life；The 1th week follow-up assessment instruments included the Bristolv Stool Form Scale, Constipation Assessment Scale, Patient Assessment of Constipation Symptoms, Visual Scale Analog, Beck Anxiety Inventory and Beck Depression Inventory II.
6. Statistical analysis Data were analyzed using SPSS 26.0 for Windows (IBM, Chicago, IL, USA). continuous variables are reported as means and standard deviations (SD), and categorical variables are reported as the number of samples and percentages. Homogeneity was tested by the Chi-square test and independent t test. Intervention effects on outcomes between the groups across repeated measurement times were analyzed by the linear mixed model using an exchangeable working correlation structure and time treated as a categorical variable that was represented by two dummy-coded variables. This study a value of p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) functional classes I-III
* Constipation(had fewer than three bowel movements a week)
* Conscious clear and communicable

Exclusion Criteria:

* Other serious diseases
* Wounds or infections in both ears

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline constipation at 2 weeks by using the Bristolv Stool Form Scale | baseline, Weeks 1 and 2
  Outcomes were assessed by using the Bristolv Stool Form Scale. This scale categorized tools between type 1 (hard lumps) and type 7 (watery diaphragm). Type 1 was separate hard lump like nuts(hard to pass), type 2 was sausage-shaped but lumpy, type 3 was like a sausage but with cracks on its surface, type 4 was like a sausage or snake, smooth and soft, type 5 was soft blobs with clear-cut edges (passed easily), type 6 is fluffy pieces with ragged edges (a mushy stool), and type 7 was watery, no solid pieces (entirely liquid). Stool types were then classified based on the Rome III criteria as stool types 1 and 2 as constipation, types 3, 4, and 5 as normal stool form, and types 6 and 7 as diarrhea,
Change from Baseline constipation at 2 weeks by using the Constipation Assessment Scale | baseline, Weeks 1 and 2
  Outcomes were assessed by using the Constipation Assessment Scale. The CAS comprised of 8 items, and each item used a 3-point Likert-type scale ranging 0~2, with a total score of 0 to 16. A higher score indicated severer constipation symptom.
Change from Baseline constipation at 2 weeks by using the Visual Scale Analog for constipation | baseline, Weeks 1 and 2
  Outcomes were assessed by using the Visual Scale Analog for constipation. The VSAQ was used to measure the immediate severity of constipation, with a 10 cm straight line with 0 on the far left (0 score) and 10 cm (10 scores) on the far right. A score ≥ 3 indicated constipation, a higher score indicating severer constipation,
Change from Baseline constipation at 2 weeks by using the Patient Assessment of Constipation Symptoms . | baseline, Weeks 1 and 2
  Outcomes were assessed by using the Patient Assessment of Constipation Symptoms .This scale comprised of 12 items with 3 subscales, including stool symptoms, rectal symptoms, and abdominal symptoms. Each item used a 5-point Likert-type scale ranging 0~4, with a total score of 0 to 48. A higher score indicated symptom severity.

SECONDARY OUTCOMES:
Change from Baseline Body constitution in Chinese Medicine at 2 weeks | at baseline, Weeks 2
  Outcomes were assessed by using the Constitution in Chinese Medicine Questionnaire. It consisted of 60 items and categorized into 9 subscales, including yang-deficient (7 items), yin-deficient (8 items), qi-deficient (8 items), phlegm-dampness (8 items), damp-heat (6 items), stagnant blood (7 items), inherited special (7 items), stagnant qi (7 items), and balanced (8 items). The items were on a 5-point Likert scale, with high scores indicating a higher likelihood of having the given body constitution. A threshold of 30 or higher points on a subscale was used to classify having that body constitution.
Change from Baseline Anxiety at 2 weeks | at baseline, Weeks 1 and 2
  Outcomes were assessed by using the Beck Anxiety Inventory. This scale consisted of 21 items that used a 4-point Likert-type scale ranging 0~3, with a total score of 0 to 63. The normal score range was 0-16, 17-22 for mild anxiety, 23-30 for moderate anxiety , and 31-63 for severe anxiety.
Change from Baseline Depression at 2 weeks | at baseline, Weeks 1 and 2
  Outcomes were assessed by using the Beck Depression Inventory II. This scale consisted of 21 items that used a 4-point Likert-type scale ranging 0~3, with a total score of 0 to 63. The normal score range was 0-16, 17-22 for mild depression, 23-30 for moderate depression, and 31-63 for severe depression.
Patient Assessment of Constipation Quality of Life | at baseline, Weeks 2
  Outcomes were assessed by using the Patient Assessment of Constipation Quality of Life, constipation affecting in daily life. It comprised of 28 items with 4 subscales, including worries and concerns, physical discomfort, psychosocial discomfort, and satisfaction. Each item used a 5-point Likert-type scale ranging 0~4, with a total score of 0 to 112. A lower score indicated better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ting Chen, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No